CLINICAL TRIAL: NCT03736135
Title: Cortisol Levels as a Measure of Accumulated Physiological Stress in Mechanical Ventilated ICU Patients: the Relationship With Premorbid Frailty, Functional, Cognitive and Psychopathological Impairment in the ICU Survivors
Brief Title: Cortisol Levels as a Measure of Accumulated Physiological Stress in ICU Patients Undergoing Mechanical Ventilation
Acronym: Corti-COG
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Sol Fernandez-Gonzalo, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CIR2017/032
Record Dates: First submitted 2018-10-22; First posted 2018-11-08 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Critical Illness
Keywords: Cortisol; Post-ICU syndrome; Cognitive impairment; Anxiety and depressive symptoms; Mechanical ventilated patients
MeSH Terms: conditions — Critical Illness; Cognitive Dysfunction; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critical illness is a situation of severe and prolonged stress for patients with mechanical ventilation (MV). Between 40-80% of these patients present the Post-ICU syndrome, a set of physical, cognitive, psychological alterations at hospital discharge. In more than a third of the ICU survivors, these sequelae become chronic being observed months and even years after ICU stay.

The characteristics of the Post-ICU syndrome have been related to different risk factors associated with the critical illness and its management. However, the impact of accumulated physiological stress is still unknown. The physiological response to prolonged stress generates high levels of cortisol that have been related to the loss of muscle tissue, cognitive and psychological alterations in both clinical populations and healthy subjects. The concentration of cortisol in plasma is not a measure of adequate physiological stress due to the dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis during critical illness. Therefore, the objective of this study is to assess the levels of accumulated cortisol in human hair (CHH) during the different stages of the critical illness and its recovery, as well as to explore its relationship with the functional and neuropsychological sequelae observed in the ICU survivors.

DETAILED DESCRIPTION:
A prospective pilot study has been proposed in 50 critical patients with> 24 hours of mechanical ventilation. CHH levels will be recorded at admission, 1 month and 1 year after ICU discharge. In all survivors, the presence of delirium will be assessed during the ICU stay and the functional, cognitive and psychological status will be assessed at short (1 month after ICU discharge) and long term (1 year after ICU discharge).

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with >24hours of mechanical ventilation

Exclusion Criteria:

* Previous neurological and/or psychiatric pathology
* Sensory alterations that prevent the application of the neurocognitive tests
* Cognitive impairment prior to ICU admission (Score >57 in the Short Form of the Informant Questionnaire on Cognitive. Decline -Short IQCODE-)
* Sever alopecia
* Rejection of voluntary participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients undergoing mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Accumulated physiological stress | At admission
  Levels of Cortisol in Human Hair (CHH)
Accumulated physiological stress | 1 month after discharge
  Levels of Cortisol in Human Hair (CHH)
Accumulated physiological stress | 1 year after discharge
  Levels of Cortisol in Human Hair (CHH)

SECONDARY OUTCOMES:
Delirium | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 3 months
  Confusion Assessment Method for ICU(CAM-ICU)
Comorbidity index | At ICU admission
  Charlson comorbidity index
Frailty index | At ICU admission
  Clinical frailty scale of Rockwood (Range 1 to 9 from 'Very fit patient' to ' Terminally ill patient'
Post-ICU syndrome physical sequelae | 1 month after discharge
  Functional score (Muscle weakness - Grip strength)
Post-ICU syndrome physical sequelae | 1 year after discharge
  Functional score (Muscle weakness - Grip strength)
Post-ICU syndrome functional sequelae | 1 month after discharge
  Functional score (Functional Morbidity - Time Up&Go)
Post-ICU syndrome functional sequelae | 1 year after discharge
  Functional score (Functional Morbidity - Time Up&Go)
Post-ICU syndrome cognitive sequelae | 1 month after discharge
  Neurocognitive score (Neurocognitive Indexes based in the neuropsychological tests)
Post-ICU syndrome cognitive sequelae | 1 year after discharge
  Neurocognitive score (Neurocognitive Indexes based in the neuropsychological tests)
Post-ICU syndrome psychological sequelae | 1 month after discharge
  Psicological status (Anxiety & Depression score)
Post-ICU syndrome psychological sequelae | 1year after discharge
  Psicological status (Anxiety & Depression score)

OTHER OUTCOMES:
Illness severity | At ICU admission
  Acute Physiology and Chronic Health Evaluation (APACHE II)
Days of MV | From date of intubation in ICU until the date of extubation in ICU or date of death from any cause, whichever came first, assessed up to 3 months
  Time with mechanical ventilation
ICU stay | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 24 months
  Days in ICU
Hospital stay | From date of ICU discharge until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 24 months
  Days in hospital after ICU discharge
Level of f alertness or agitation | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 3 months
  Richmond Agitation-Sedation Scale (RASS)
Dosis of sedatives and opioids | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 3 months
  Daily accumulated dosis of sedatives and opioids

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Blanch, PhD, Study Director — I3PT-Fundació Parc Taulí
Locations (1):
- Fundacio Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Berghe GV. Novel insights in the HPA-axis during critical illness. Acta Clin Belg. 2014 Dec;69(6):397-406. doi: 10.1179/2295333714Y.0000000093. PMID 25409903
- [Background] Cuesta JM, Singer M. The stress response and critical illness: a review. Crit Care Med. 2012 Dec;40(12):3283-9. doi: 10.1097/CCM.0b013e31826567eb. PMID 22975887
- [Background] Karnatovskaia LV, Johnson MM, Benzo RP, Gajic O. The spectrum of psychocognitive morbidity in the critically ill: a review of the literature and call for improvement. J Crit Care. 2015 Feb;30(1):130-7. doi: 10.1016/j.jcrc.2014.09.024. Epub 2014 Oct 2. PMID 25449881
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Hopkins RO. The brain after critical illness: effect of illness and aging on cognitive function. Crit Care. 2013 Feb 6;17(1):116. doi: 10.1186/cc11913. PMID 23384320
- [Background] Jackson JC, Hart RP, Gordon SM, Shintani A, Truman B, May L, Ely EW. Six-month neuropsychological outcome of medical intensive care unit patients. Crit Care Med. 2003 Apr;31(4):1226-34. doi: 10.1097/01.CCM.0000059996.30263.94. PMID 12682497
- [Background] Reser JE. Chronic stress, cortical plasticity and neuroecology. Behav Processes. 2016 Aug;129:105-115. doi: 10.1016/j.beproc.2016.06.010. Epub 2016 Jun 19. PMID 27334119
- [Background] Liston C, Miller MM, Goldwater DS, Radley JJ, Rocher AB, Hof PR, Morrison JH, McEwen BS. Stress-induced alterations in prefrontal cortical dendritic morphology predict selective impairments in perceptual attentional set-shifting. J Neurosci. 2006 Jul 26;26(30):7870-4. doi: 10.1523/JNEUROSCI.1184-06.2006. PMID 16870732
- [Background] Allen AP, Curran EA, Duggan A, Cryan JF, Chorcorain AN, Dinan TG, Molloy DW, Kearney PM, Clarke G. A systematic review of the psychobiological burden of informal caregiving for patients with dementia: Focus on cognitive and biological markers of chronic stress. Neurosci Biobehav Rev. 2017 Feb;73:123-164. doi: 10.1016/j.neubiorev.2016.12.006. Epub 2016 Dec 13. PMID 27986469
- [Background] Hermans G, De Jonghe B, Bruyninckx F, Van den Berghe G. Clinical review: Critical illness polyneuropathy and myopathy. Crit Care. 2008;12(6):238. doi: 10.1186/cc7100. Epub 2008 Nov 25. PMID 19040777
- [Background] Boonen E, Vervenne H, Meersseman P, Andrew R, Mortier L, Declercq PE, Vanwijngaerden YM, Spriet I, Wouters PJ, Vander Perre S, Langouche L, Vanhorebeek I, Walker BR, Van den Berghe G. Reduced cortisol metabolism during critical illness. N Engl J Med. 2013 Apr 18;368(16):1477-88. doi: 10.1056/NEJMoa1214969. Epub 2013 Mar 19. PMID 23506003
- [Background] Stalder T, Kirschbaum C. Analysis of cortisol in hair--state of the art and future directions. Brain Behav Immun. 2012 Oct;26(7):1019-29. doi: 10.1016/j.bbi.2012.02.002. Epub 2012 Feb 15. PMID 22366690
- [Background] McLennan SN, Ihle A, Steudte-Schmiedgen S, Kirschbaum C, Kliegel M. Hair cortisol and cognitive performance in working age adults. Psychoneuroendocrinology. 2016 May;67:100-3. doi: 10.1016/j.psyneuen.2016.01.029. Epub 2016 Feb 1. PMID 26881835